CLINICAL TRIAL: NCT05188976
Title: Validity Assessment of End-tidal Carbon Dioxide Levels in Respiratory Disease
Brief Title: Assessment of End-tidal Carbon Dioxide Levels in Respiratory Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Hospital Organization Minami Kyoto Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-31
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Disease
Keywords: PetCO2
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood gas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to evaluate the correlation between PetCO2, PaCO2, and PtcCO2 in patients with respiratory diseases. The investigators also evaluate the correlation between PetCO2, PaCO2, and PtcCO2 changes over time.

DETAILED DESCRIPTION:
Partial pressure of carbon dioxide(PCO2) is mainly evaluated by partial pressure of arterial carbon dioxide (PaCO2), and is used as an index for prognosis and NPPV introduction in chronic respiratory failure. Arterial blood gas analysis for PaCO2 measurement is the most accurate test value, but it is invasive and frequent tests are difficult and cannot be performed at home. The transcutaneous PCO2 (PtcCO2) is a non-invasive measurement and its measured value is close to PaCO2, and it can be measured continuously, which is useful for monitoring patients with chronic respiratory failure. However, PtcCo2 has not been applied at home due to technical problems (necessity of calibration, periodic drift, etc.). The end-tidal pressure of expired CO2 (PetCO2) can be measured non-invasively, easily and continuously. PetCO2 is mainly used for patients undergoing mechanical ventilation, and its accuracy and stability have been evaluated. The investigators decided to investigate whether PetCO2 is useful for monitoring respiratory status in patients with respiratory disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with respiratory disorder.
* Subjects who are clinically stable for the last 2 weeks

Exclusion Criteria:

* Subjects who required treatment with antibacterial agents or oral/intravenous steroids for pneumonia or exacerbation of respiratory disease in the last 2 weeks.
* Subjects with severe complications such as cardiovascular disease, liver disease, renal disease, and neurological disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with respiratory disease such as COPD, IP
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between PetCO2, PaCO2, and PtcCO2 | One to three months

SECONDARY OUTCOMES:
Correlation of changes over time between PetCO2, PaCO2 , and PtcCO2 | One to three months
Relationship between PetCO2 and respiratory symptoms evaluated by The COPD Assessment Test (CAT) and mMRC (modified British Medical Research Council) | One to three months

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto, Japan